CLINICAL TRIAL: NCT03034122
Title: Is Caffeine an Environmental Modifier in Huntington's Disease?
Acronym: CrEAM-HD
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2015_67; 2016-A00892-49 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2017-01-24; First posted 2017-01-27 (Estimated); Last update posted 2025-12-23 (Actual); Status verified 2024-12

CONDITIONS: Huntington Disease
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of the study is to establish if caffeine consumption is associated with the evolution of the disease in premanifest HD.

ELIGIBILITY:
Inclusion Criteria:

* HD mutation carriers (>36 CAG)
* premanifest (total motor UHDRS < 5)
* estimated time to diagnosis between 3 and 10 years
* adults older than 21 years (in order to exclude juvenile patients who begin the disease before 21 years)
* informed consent signed
* with a social protection

Exclusion Criteria:

* MRI contraindication
* pregnant and lactating women
* People under guardianship, trusteeship, deprive of freedom

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: premanifest HD subjects
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-04-12 (Actual)

PRIMARY OUTCOMES:
Change in striatal volume | at 2 years

SECONDARY OUTCOMES:
Unified Huntington's Disease Rating Scale (UHDRS) | at 1 years, at 2 years
  measure the change of motor scale for exposure caffeine groups
SDMT -symbol digit modality test | at 1 years, at 2 years
  measure the change of cognitive score for exposure caffeine groups
Stroop test | at 1 years, at 2 years
  measure the change of cognitive score for exposure caffeine groups
PBA (problem behaviors assessment) | at 1 years, at 2 years
  the PBA is a semi structured clinical interview measuring the presence, severity and frequency of 11 key behavioural symptoms.
  measure the change score and subscores for apathy, obsessive-compulsive disorders, irritability, anxiety and depression,
score at Epworth sleepiness scale | at 1 years, at 2 years
  measure the change of sleepiness scale for exposure caffeine groups
MRI | at 1 years, at 2 years
  measure the change of image of the whole brain and other deep gray nuclei atrophy

CONTACTS AND LOCATIONS:
Overall Officials: Clémence Simonin, MD, Principal Investigator — University Hospital, Lille
Locations (10):
- France (10):
  - CHU de Amiens, Amiens
  - CHU de Angers, Angers
  - CHU Pellegrin, Bordeaux
  - CHU de Grenoble, Grenoble
  - Hôpital Roger Salengro, CHRU, Lille
  - CHU Montpellier, Montpellier
  - CHU de Nancy, Nancy
  - AH-HP La Pitié-Salpétrière, Paris
  - AH-HP, Hôpital Henri Mondor, Paris
  - CHU Purpan, Toulouse

IPD SHARING:
Plan to Share IPD: No